CLINICAL TRIAL: NCT04129541
Title: Same-day Discharge After Reconstructive Pelvic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000026647
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Reconstructive Pelvic Surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDD (Active Comparator): Patients will receive routine care during their admission for surgery. A standard voiding trial will be performed in the PACU for all patients. Patients in the planned same day discharge (SDD) cohort will be discharged from the PACU once they meet standard discharge criteria.
  Interventions: Other: Same Day Discharge
- OH (Active Comparator): Patients will receive routine care during their admission for surgery. A standard voiding trial will be performed in the PACU for all patients. Patients in the planned overnight hospitalization (OH) group will be discharged on post-operative day 1 once they meet standard discharge criteria.
  Interventions: Other: Overnight Hospitalization

INTERVENTIONS:
Other: Same Day Discharge — Patients in the planned same day discharge (SDD) cohort will be discharged from the PACU once they meet standard discharge criteria.
  Arms: SDD
Other: Overnight Hospitalization — Patients in the planned overnight hospitalization (OH) group will be discharged on post-operative day 1 once they meet standard discharge criteria.
  Arms: OH

SUMMARY:
The purpose of this study is to determine the safety and acceptability of same-day discharge after surgery for pelvic floor disorders. The study hypotheses are that same-day discharge after reconstructive pelvic surgery is safe and improves patient satisfaction when compared to overnight hospitalization.

DETAILED DESCRIPTION:
This study is a randomized clinical trial comparing same day discharge and overnight hospitalization after reconstructive pelvic surgery. Patients who are scheduled to undergo surgery for pelvic organ prolapse (POP) and/or stress urinary incontinence (SUI) will be recruited at their preoperative visit. Patients will be counseled regarding the existing evidence demonstrating the safety of same day discharge after hysterectomy and pelvic floor reconstructive surgery. Eligible patients who provide consent will be randomized to same day discharge or overnight hospitalization following surgery.

Patients will receive routine care during their admission for surgery. A standard voiding trial will be performed in the Post-Anesthesia Care Unit (PACU) for all patients. Patients in the planned same day discharge (SDD) cohort will be discharged from the PACU once they meet standard discharge criteria. If the patients require unplanned hospitalization (UH), the reason for hospitalization will be noted. Patients in the planned overnight hospitalization (OH) group will be discharged on post-operative day 1 once they meet standard discharge criteria.

At their postoperative office visit, all patients will complete surveys evaluating patient satisfaction. Demographic, surgical, and hospital admission data will be collected from the medical record. Information will also be collected regarding any complications, emergency department (ED) visits, unplanned office visits, readmissions, and reoperations within 8 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for pelvic organ prolapse, with or without concomitant hysterectomy or incontinence procedure.

Exclusion Criteria:

* Patients undergoing concomitant non-gynecologic procedure
* The presence of: gynecologic malignancy, American Society of Anesthesiologists (ASA) class >2, severe cardiovascular or pulmonary comorbidities, prior anesthesia complication, or obstructive sleep apnea
* Anyone living alone with no family/friend/caretaker to assist the patient on day of surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Recovery Score | 6 to 8 weeks after surgery
  Quality of recovery will be assessed using the Quality of Recovery-15 (QoR-15) at baseline, 48 hours postop, and 6-8 weeks postop. The QoR-15 consists of 15 questions scored on a 0 to 10 scale, maximum score 150. Higher scores indicate good recovery after surgery while lower scores indicate poor recovery.
Patient Satisfaction | 6 to 8 weeks after surgery
  Patient satisfaction will be assessed using the Patient Global Impression of Improvement (PGI-I) at 6-8 weeks postop. The PGI-I consists of 1 question scored 1-7, with lower number indicating better global improvement.

SECONDARY OUTCOMES:
Safety Measures: frequency of post operative complications | Up to 8 weeks after surgery
  Safety will be measured by the frequency of post operative complications, this will include counts of emergency department visits, readmissions, and reoperations; as well as frequency of any unplanned office visits and phone calls within 8 weeks after surgery.
Quality of Recovery (baseline) | Baseline
  Quality of recovery will be assessed using the Quality of Recovery-15 (QoR-15) at baseline, 48 hours postop, and 6-8 weeks postop. The QoR-15 consists of 15 questions scored on a 0 to 10 scale, maximum score 150. Higher scores indicate good recovery after surgery while lower scores indicate poor recovery.
Quality of Recovery (48 hours) | 48 hours postop
  Quality of recovery will be assessed using the Quality of Recovery-15 (QoR-15) at baseline, 48 hours postop, and 6-8 weeks postop. The QoR-15 consists of 15 questions scored on a 0 to 10 scale, maximum score 150. Higher scores indicate good recovery after surgery while lower scores indicate poor recovery.
Quality of Recovery (at postop visit) | 48 hours postop
  Quality of recovery will be assessed using the Quality of Recovery-15 (QoR-15) at baseline, 48 hours postop, and 6-8 weeks postop. The QoR-15 consists of 15 questions scored on a 0 to 10 scale, maximum score 150. Higher scores indicate good recovery after surgery while lower scores indicate poor recovery.
Pelvic Floor Distress (baseline) | Baseline
  Pelvic floor distress will be assessed using the Pelvic Floor Distress Inventory (PFDI-20) summary score at baseline and 6-8 weeks postop. The PFDI-20 consists of 20 questions scored on a 0 to 4 scale, divided into three scales consisting of 6, 8, and 6 questions each. For scoring, the mean value is obtained for each scale (0-4) and multiplied by 25 to obtain the scale score (0-100). The summary PFDI score is the sum of the three scale scores (0-300). Higher score indicates higher distress from pelvic floor disorder symptoms.
Pelvic Floor Distress (postop) | 6 to 8 weeks after surgery
  Pelvic floor distress will be assessed using the Pelvic Floor Distress Inventory (PFDI-20) summary score at baseline and 6-8 weeks postop. The PFDI-20 consists of 20 questions scored on a 0 to 4 scale, divided into three scales consisting of 6, 8, and 6 questions each. For scoring, the mean value is obtained for each scale (0-4) and multiplied by 25 to obtain the scale score (0-100). The summary PFDI score is the sum of the three scale scores (0-300). Higher score indicates higher distress from pelvic floor disorder symptoms.
Pelvic Floor Impact (baseline) | Baseline
  Pelvic floor impact will be assessed using the Pelvic Floor Impact Questionnaire (PFIQ-7) at baseline and 6-8 weeks postop. The PFIQ-7 consists of 21 questions scored on a 0 to 3 scale, divided into three scales consisting of 7 questions each. For scoring, the mean value is obtained for each scale (0-3) and multiplied by 100/3 to obtain the scale score (0-100). The summary PFIQ score is the sum of the three scale scores (0-300). Higher score indicates higher impact of pelvic floor disorders on activities, relationships, and feelings.
Pelvic Floor Impact (postop) | 6 to 8 weeks after surgery
  Pelvic floor impact will be assessed using the Pelvic Floor Impact Questionnaire (PFIQ-7) at baseline and 6-8 weeks postop. The PFIQ-7 consists of 21 questions scored on a 0 to 3 scale, divided into three scales consisting of 7 questions each. For scoring, the mean value is obtained for each scale (0-3) and multiplied by 100/3 to obtain the scale score (0-100). The summary PFIQ score is the sum of the three scale scores (0-300). Higher score indicates higher impact of pelvic floor disorders on activities, relationships, and feelings.

CONTACTS AND LOCATIONS:
Overall Officials: Oz Harmanli, MD, Principal Investigator — Chief, Yale Urogynecology and Pelvic Reconstructive Surgery

IPD SHARING:
Plan to Share IPD: No